CLINICAL TRIAL: NCT07133256
Title: Effects of Aerobic Versus Resistance Training on Bone Metabolism in Stage 3-4 Chronic Kidney Disease: A Randomized Controlled Trial
Brief Title: Effects of Aerobic Versus Resistance Training on Bone Metabolism in Stage 3-4 Chronic Kidney Disease
Acronym: CKD-BONE-EX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, lecturer, Sinai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU.REC.2025(45H)
Record Dates: First submitted 2025-08-06; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Osteopenia; Bone Metabolism Disorders; Chronic Kidney Disease (Stage 3-4); Mineral and Bone Disorder (CKD-MBD)
Keywords: Chronic kidney disease; RANKL, OPG/RANKL Ratio; Osteoprotegerin; Aerobic Exercise; Resistance Exercise; Bone mineral density
MeSH Terms: conditions — Bone Diseases, Metabolic; Renal Insufficiency, Chronic; Calcinosis; Bone Diseases; Chronic Kidney Disease-Mineral and Bone Disorder; Osteopetrosis, mild autosomal recessive form | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Interventional (Clinical Trial)
Who Masked: Outcomes Assessor
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Exercise Group (Group A) (Experimental): Participants in this arm engaged in supervised resistance training three times per week for six months. Each session included:
  5-minute warm-up with dynamic stretching and range-of-motion exercises
  30-minute resistance training using weight machines targeting major muscle groups (upper limbs, lower limbs, and trunk)
  Intensity: 60% to 80% of one-repetition maximum (1-RM), adjusted progressively
  10-minute cool-down with static stretching Sessions were monitored by trained physiotherapists.
  Interventions: Behavioral: Resistance Exercise
- Aerobic Exercise Group (Group B) (Active Comparator): Participants in this arm performed supervised aerobic exercise (treadmill walking) three times per week for six months. Each session included:
  5-minute warm-up
  30-minute treadmill walking at 60%-80% of age-predicted maximum heart rate (HRmax = 220 - age)
  10-minute cool-down Exercise sessions were supervised by trained exercise professionals and tailored to maintain target heart rate zones.
  Interventions: Behavioral: Aerobic Training

INTERVENTIONS:
Behavioral: Resistance Exercise — Structured machine-based resistance exercise protocol performed under supervision, targeting osteogenic loading to improve bone mineral density and alter bone metabolism markers in CKD stage 3-4 patients.
  Arms: Resistance Exercise Group (Group A)
Behavioral: Aerobic Training — Participants in this arm performed supervised aerobic exercise (treadmill walking) three times per week for six months. Each session included:
  5-minute warm-up
  30-minute treadmill walking at 60%-80% of age-predicted maximum heart rate (HRmax = 220 - age)
  10-minute cool-down Exercise sessions were supervised by trained exercise professionals and tailored to maintain target heart rate zones.
  Arms: Aerobic Exercise Group (Group B)

SUMMARY:
This randomized controlled trial investigates the comparative effects of aerobic versus resistance training on bone mineral density (BMD) and bone metabolism markers in patients with stage 3 or 4 chronic kidney disease (CKD). The primary aim is to evaluate the impact of two distinct exercise modalities on serum osteoprotegerin (OPG), receptor activator of nuclear factor kappa-B ligand (RANKL), and the OPG/RANKL ratio, as well as densitometric changes at key skeletal sites.

DETAILED DESCRIPTION:
Chronic kidney disease-mineral and bone disorder (CKD-MBD) is a common complication in non-dialysis CKD patients, driven by disrupted calcium-phosphate metabolism, secondary hyperparathyroidism, and altered bone remodeling pathways, such as the OPG-RANKL axis. Exercise is an emerging non-pharmacological strategy to mitigate skeletal deterioration in CKD, yet the differential effects of aerobic and resistance training on bone health remain poorly understood in this population.

This study recruited 60 CKD patients (stage 3-4, aged 30-50 years) and randomly allocated them into two groups (n=30 each): a resistance training group and an aerobic exercise group. Both groups underwent supervised exercise 3 times per week for six months. Bone mineral density was assessed using dual-energy X-ray absorptiometry (DEXA) at the lumbar spine (L2-L4), femoral neck, and distal radius. Serum concentrations of OPG and RANKL were measured via ELISA at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30 to 50 years
* Diagnosed with stage 3 or 4 chronic kidney disease (non-dialysis dependent)
* BMI between 20 and 24 kg/m²
* Not currently taking medications that affect bone density (e.g., corticosteroids, bisphosphonates)
* Non-smokers and abstinent from alcohol
* Not receiving hormone replacement therapy
* Willing and able to participate in supervised exercise sessions for 6 months

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus
* Uncontrolled hypertension
* History of cardiovascular, musculoskeletal, endocrine, or metabolic bone disease
* Pregnant or planning pregnancy during the study period
* Participation in a structured exercise program within the last 3 months
* Contraindications to exercise as determined by medical evaluation
* Use of investigational drugs or enrollment in another clinical trial during the study period

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 30 to 50
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Change in Serum Osteoprotegerin (OPG) and RANKL Concentrations | Baseline to 6 months post-intervention
  To determine biochemical changes in bone metabolism markers. Both OPG (pg/mL) and RANKL (ng/mL) are measured using validated ELISA kits.
Change in Bone Mineral Density (BMD) | Baseline to 6 months post-intervention
  To assess densitometric changes in skeletal structure due to exercise. BMD is measured in g/cm² using ISCD-certified DEXA equipment.
Change in OPG/RANKL Ratio | To assess the regulatory balance of bone remodeling. A higher OPG/RANKL ratio reflects reduced osteoclastic activity and improved bone metabolic status.
  Baseline to 6 months post-intervention

SECONDARY OUTCOMES:
Change in eGFR (estimated Glomerular Filtration Rate) | Baseline to 6 months
  To explore the potential renal benefits of structured exercise in CKD patients. Measured in mL/min/1.73 m².
Change in Serum Albumin and Hemoglobin Levels | Baseline to 6 months
  These indicators provide information about overall nutritional and hematologic status. Albumin (g/dL) and Hemoglobin (g/dL) are assessed via standard lab procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shehab Abd E-Kader, Professor, Principal Investigator — 1Department of Physical Therapy, Faculty of Medical Rehabilitation Sciences, King Abdulaziz University, Jeddah, Saudi Arabia.
Locations (1):
- Manshyet El-Bakry Hospital, Cairo, Egypt